CLINICAL TRIAL: NCT04278144
Title: Phase 1/2 Study of BDC-1001 as a Single Agent and in Combination With Nivolumab in Patients With Advanced HER2-Expressing Solid Tumors
Brief Title: A First-in-human Study Using BDC-1001 as a Single Agent and in Combination With Nivolumab in Advanced HER2-Expressing Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Bolt Biotherapeutics, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI-20201001
Record Dates: First submitted 2020-02-12; First posted 2020-02-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HER2-positive Solid Tumors; HER2-positive Breast Cancer; HER2-positive Colorectal Cancer; HER2-positive Gastroesophageal Cancer; HER2-positive Endometrial Cancer
Keywords: HER2; ERBB2; Immunotherapy; Gastric Cancer; Gastroesophageal junction; Breast Cancer; Stomach Cancer; Colorectal Cancer; Gastrointestinal Cancer; Non-Small Cell Lung Cancer; Biliary Tract Cancer; Head and Neck Cancer; Urothelial Cancer; Endometrial Cancer; TLR7/8 agonist
MeSH Terms: conditions — Stomach Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms; Head and Neck Neoplasms; Endometrial Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Multiple ascending dose and dose-expansion of BDC-1001 administered as a single agent or in combination with nivolumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single agent BDC-1001 (Experimental): Escalating doses followed by expansion targeting HER2-expressing advanced malignancies
  Interventions: Drug: BDC-1001
- Combination BDC-1001 plus nivolumab (Experimental): Escalating doses followed by expansion targeting HER2-expressing advanced malignancies
  Interventions: Drug: BDC-1001; Drug: Nivolumab

INTERVENTIONS:
Drug: BDC-1001 — Immune stimulating antibody conjugate (ISAC), consisting of an anti-HER2 monoclonal antibody conjugated to a TLR 7/8 dual agonist
Drug: Nivolumab — Programmed death receptor-1 (PD 1)-blocking antibody
  Other Names: Opdivo
  Arms: Combination BDC-1001 plus nivolumab

SUMMARY:
A first-in-human study using BDC-1001 as a single agent and in combination with nivolumab in HER2 expressing advanced malignancies

DETAILED DESCRIPTION:
This study has four parts. Part 1 is a dose escalation of BDC-1001 as a single agent to determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), or maximum protocol dose (MPD) recommended for Part 3. In Part 3, the selected dose will be administered as monotherapy to patients with selected advanced malignancies. Part 2 is a dose escalation of BDC-1001 in combination with nivolumab to determine the maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), or maximum protocol dose (MPD) recommended for Part 4. In Part 4, the selected dose will be administered in combination with nivolumab to patients with selected advanced malignancies.

Bolt amended the protocol to transition any subjects still receiving BDC-1001 to continue receiving BDC-1001 in the Maintenance Phase. Subjects remaining on BDC-1001 will continue to receive BDC-1001 until a criterion for discontinuation has been met.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient must have an advanced solid tumor with documented HER2-protein expression or gene amplification for which approved therapies have been exhausted or are not clinically indicated.
* Measurable disease as determined by RECIST v.1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Tumor tissue (archival or collected prior to the study start) available for exploratory biomarker evaluation.

Key Exclusion Criteria:

* History of severe hypersensitivity to any ingredient of the study drug(s), including trastuzumab or other monoclonal antibody.
* Previous treatment with a TLR 7, TLR 8 or a TLR 7/8 agonist.
* Impaired cardiac function or history of clinically significant cardiac disease
* Human Immunodeficiency virus (HIV) infection, active hepatitis B infection, or hepatitis C infection.
* Active SARS-CoV-2 infection
* Untreated central nervous system (CNS), epidural tumor or metastasis, or brain metastasis.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 2 years
  Escalation period
Incidence and nature of dose-limiting toxicities (DLTs) | up to 21 days
  Escalation period
Incidence of potential-immune related toxicities | 2 years
  Escalation period
Maximum tolerable dose (MTD) or a tolerated dose below MTD | 2 years
  Escalation period
Objective response rate (ORR) of confirmed complete or partial responses (CR, PR) | 2 years
  Expansion period

SECONDARY OUTCOMES:
PK (Cmax) of BDC-1001 | 2 years
  Escalation and expansion periods
PK (Cmin) of BDC-1001 | 2 years
  Escalation and expansion periods
PK (AUC0-t) of BDC-1001 | 2 years
  Escalation period
PK (AUC0-inf) of BDC-1001 | 2 years
  Escalation period
PK (CL) of BDC-1001 | 2 years
  Escalation period
PK (Vz) of BDC-1001 | 2 years
  Escalation period
PK (t1/2) of BDC-1001 | 2 years
  Escalation period
Objective response rate (ORR) using RECIST 1.1 | 2 years
  Escalation period
Duration of response (DOR) | 2 years
  Escalation and expansion periods
Disease control rate (DCR) of confirmed CR, PR, or stable disease (SD) lasting 4 or more weeks | 2 years
  Escalation and expansion periods
Progression Free Survival (PFS) | 2 years
  Escalation and expansion periods
Incidence of anti-BDC-1001 antibodies | 2 years
  Escalation and expansion periods
Incidence of adverse events (AEs) and serious adverse events (SAEs) | 2 years
  Expansion period
Incidence of potential-immune related toxicities | 2 years
  Expansion period

CONTACTS AND LOCATIONS:
Overall Officials: Bolt Clinical Development, Study Director — Bolt Biotherapeutics
Locations (21):
- United States (11):
  - Stanford University, Palo Alto, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The University of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- France (3):
  - Institut Bergonie, Bordeaux
  - Institut Paoli Calmettes, Marseille
  - Institut Gustave Roussy, Villejuif
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, Seoul, Songpa-gu
- Spain (4):
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Universitario Vall d'Hebron, Barcelona, Catalonia
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No